CLINICAL TRIAL: NCT04592887
Title: Feasibility Study of FLASH Radiotherapy for the Treatment of Symptomatic Bone Metastases
Acronym: FAST-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAR-2019-02
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Bone Metastasis
Keywords: FLASH radiotherapy; Radiation treatment; Proton; Bone metastasis; Feasibility study; Pain relief; Toxicities; Extremities

STUDY DESIGN:
Intervention Model Description: Open label, single arm prospective feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- FLASH radiotherapy for painful bone metastasis(-es) (Experimental)
  Interventions: Radiation: FLASH Radiotherapy

INTERVENTIONS:
Radiation: FLASH Radiotherapy — FLASH radiotherapy is radiation treatment delivered at ultra-high dose rates compared to conventional radiation treatment.

SUMMARY:
This purpose of this study is to assess the feasibility of FLASH radiotherapy for the palliative treatment of painful bone metastases. FLASH radiotherapy is radiation treatment delivered at ultra-high dose rates compared to conventional radiation treatment.

DETAILED DESCRIPTION:
This clinical investigation is designed to assess the workflow feasibility of FLASH radiotherapy treatment in a clinical setting, as well as the toxicities, and pain relief when used to treat bone metastasis(-es) in the extremities (excluding feet, hands, wrists). FLASH radiotherapy has been shown in preclinical studies to cause less injury to surrounding normal tissues during radiation treatment, while still having similar tumor cell killing. Patients at least 18 years of age with painful bone metastases located in the limbs will be considered for the study. These patients represent an ideal population for a feasibility study of FLASH radiotherapy as they are known to benefit from the palliative effects of radiotherapy using single dose radiation regimens of 8Gy which is what is being used in this investigation. After treatment, patients will be assessed for pain response as well as any adverse side-effects of radiation. The workflow feasibility of the treatment will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patient age at least 18 years
* Up to 3 painful bone metastasis(-es) in the extremities
* Bone metastases that can be treated using pre-defined treatment field sizes (7.5 cm x 7.5 cm; 7.5 cm x 10 cm; 7.5 cm x 12 cm; 7.5 cm x 14 cm; 7.5 cm x 16 cm; 7.5 cm x 18 cm; 7.5 cm x 20 cm), without overlap of radiation fields
* Life expectancy of >2 months (in the judgement of the investigator)
* Patients who are able to comply with the protocol
* Provision of signed and dated informed consent form

Exclusion Criteria:

* Prior radiotherapy to the treatment site(s)
* Lesions of the feet, hands, wrists are not eligible treatment sites for FLASH
* More than 3 painful bone metastases of the limbs requiring palliative radiotherapy
* Tumor lysis of >50% of the circumferential bone cortex, or other factors considered to place the subject at significant risk of pathologic fracture
* Patients with bone fractures and/or metal implants in the treatment field
* Patients who will receive cytotoxic chemotherapy within 1 week prior to or 1 week following their planned radiation treatment
* Prior local therapy modality to the treatment site(s) within 2 weeks of study enrollment
* Patients with pacemakers or other implanted devices at risk of malfunction during radiotherapy
* Patients with any other medical condition or laboratory value that would, at the discretion of the investigator, preclude the patient from participation in this clinical investigation
* Patients at known risk of enhanced normal tissue sensitivity to radiotherapy due to inherited predisposition or documented comorbidity that might lead to hypersensitivity to ionizing radiation
* Patients enrolled in any other clinical studies the investigator believes to be in conflict with this clinical investigation.
* Patients who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Breneman, MD, Principal Investigator — Professor of Radiation Oncology and Neurosurgery, UCMC
Locations (1):
- Cincinnati Children's Proton Therapy Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mascia AE, Daugherty EC, Zhang Y, Lee E, Xiao Z, Sertorio M, Woo J, Backus LR, McDonald JM, McCann C, Russell K, Levine L, Sharma RA, Khuntia D, Bradley JD, Simone CB 2nd, Perentesis JP, Breneman JC. Proton FLASH Radiotherapy for the Treatment of Symptomatic Bone Metastases: The FAST-01 Nonrandomized Trial. JAMA Oncol. 2023 Jan 1;9(1):62-69. doi: 10.1001/jamaoncol.2022.5843. PMID 36273324
- [Derived] Daugherty EC, Mascia A, Zhang Y, Lee E, Xiao Z, Sertorio M, Woo J, McCann C, Russell K, Levine L, Sharma R, Khuntia D, Bradley J, Simone CB 2nd, Perentesis J, Breneman J. FLASH Radiotherapy for the Treatment of Symptomatic Bone Metastases (FAST-01): Protocol for the First Prospective Feasibility Study. JMIR Res Protoc. 2023 Jan 5;12:e41812. doi: 10.2196/41812. PMID 36206189
- [Derived] Maity A, Koumenis C. Shining a FLASHlight on Ultrahigh Dose-Rate Radiation and Possible Late Toxicity. Clin Cancer Res. 2022 Sep 1;28(17):3636-3638. doi: 10.1158/1078-0432.CCR-22-1255. PMID 35736814

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FLASH Radiotherapy for Painful Bone Metastasis(-es)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FLASH Radiotherapy for Painful Bone Metastasis(-es)
Number analyzed (Participants) | 10
Age, Customized [Count of Participants; unit: Participants] — Participant age at least 18 years
  Participants
    Participant age at least 18 year | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Workflow Feasibility
Description: Number of participants with total time on table under one hour. The investigational site staff will measure the time for participant set-up and positioning on the treatment couch, imaging and FLASH treatment delivery. The workflow feasibility outcome measure is met for an individual subject if total time on table is measured as less than one hour.
  The outcome measure data table provides the mean and full range of time on table (as measured in minutes) for the 10 participants. The participant with a treatment time of 33 minutes received treatment to two separate metastatic sites; remaining 9 participants received treatment to a single metastatic site.
Time Frame: Will be assessed on day of treatment delivery which occurs within 3 weeks of subject enrollment.
Measure: Mean (Full Range); unit: minutes
Arm/Group | FLASH Radiotherapy for Painful Bone Metastasis(-es)
Number analyzed (Participants) | 10
minutes | 15.8 [11 to 33]

2. Primary Outcome: Workflow Feasibility
Description: Number of participants whose treatment was delayed by more than 7 business days from simulation to treatment when related to the investigational device (excluding delays due to patient or facility factors not related to study treatment).
  The investigational site staff will measure the number of days delay in time to treatment due to problems involving the investigational device. The workflow feasibility outcome measure is met for an individual subject if the delay is measured as less than 7 days.
  The outcome measure data table provides the mean and full range days of treatment delay for the 10 participants.
Time Frame: Will be assessed within 4 weeks of subject enrollment.
Measure: Mean (Full Range); unit: days
Arm/Group | FLASH Radiotherapy for Painful Bone Metastasis(-es)
Number analyzed (Participants) | 10
days | 0 [0 to 0]

3. Primary Outcome: Assessment of Radiation-related Toxicities That Are Possibly, Probably, or Definitely Related to FLASH Radiotherapy.
Description: Toxicities that are possibly, probably, or definitely related to FLASH radiotherapy. Toxicities will be classified per CTCAE version 5.0.
  The outcome measure data table summarizes the total number of adverse events possibly, probably, definitely related to treatment that were reported in the 10 participant cohort. Eleven adverse events were grade 1 and one adverse event was grade 2, as classified by CTCAE version 5.0.
Time Frame: Assessed from start of treatment until subject death or lost to follow-up, up to 17.8 months
Measure: Number; unit: adverse events related to treatment
Arm/Group | FLASH Radiotherapy for Painful Bone Metastasis(-es)
Number analyzed (Participants) | 10
adverse events related to treatment
  Grade 1 adverse events | 11
  Grade 2 adverse events | 1

4. Secondary Outcome: Pain Relief
Description: Percentage of treated sites achieving pain relief as measured using patient reported outcome questionnaires (Brief Pain Inventory Questionnaire, Treated Sites Pain Questionnaire). Categories of pain relief included complete, partial, stable or progressive response.
  Complete response (CR) = no pain at 3 months Partial response (PR) = an average pain score that is ≥2 points lower than initial Stable disease (SD) = an average pain score that is ±1 point change from initial Progressive disease (PD) = an average pain score that is ≥2 points higher than initial
Time Frame: At 3 month follow up
Population: The outcome measures data table details the percentage of pain response rate (in the categories of response described above) for 12 treated sites involving 10 participants.
Measure: Number; unit: Percentage of treated sites
Units Other Than Participants: Treated Sites
Arm/Group | FLASH Radiotherapy for Painful Bone Metastasis(-es)
Number analyzed (Participants) | 10
Number analyzed (Treated Sites) | 12
Percentage of treated sites
  Complete Response | 50
  Partial Response | 16.7
  Stable Response | 25
  Progressive Reponse | 8

5. Secondary Outcome: Number of Participants Who Experienced a Pain Flare.
Description: Pain was assessed by patient reported validated 10 point pain flare questionnaire. Pain flare is defined as either of the following: A) a minimum of a two-point increase in the worst pain score for the treated site without a reduction in analgesic intake; or B) a 25% or greater increase in analgesic intake based on daily oral morphine equivalence without a reduction in the worst pain score.
Time Frame: First 10 days post FLASH treatment
Measure: Count of Participants; unit: Participants
Arm/Group | FLASH Radiotherapy for Painful Bone Metastasis(-es)
Number analyzed (Participants) | 10
Participants | 4

6. Secondary Outcome: Number of Participants With Increased Use of Pain Medication in First 10 Days Post FLASH Treatment
Description: Use of pain medication by study participant during days 1-10 following FLASH treatment was collected as it constituted one of the defining criteria (criteria B) for the pain flare outcome measure.
  Pain flare is defined as either of the following: A) a minimum of a two-point increase in the worst pain score for the treated site without a reduction in analgesic intake; or B) a 25% or greater increase in analgesic intake based on daily oral morphine equivalence without a reduction in the worst pain score.
Time Frame: Within 10 days after treatment.
Population: Four out of the 10 participants experienced a pain flare. Two of these 4 participants met criteria B) whose use of pain medication in the first 10 days after treatment met the endpoint for pain flare.
Measure: Number; unit: Participants
Arm/Group | FLASH Radiotherapy for Painful Bone Metastasis(-es)
Number analyzed (Participants) | 10
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at Day 2, 15, Months 1, 2, 3, long term, or subject death/lost to follow up, up to 17.8 months (for the longest follow up). Length of follow up for each subject is as follows: #1: 2.3 months, #2: 16.5 months, #3: 17.8 months, #4: 9.3 months, #5: 3 months, #6: 4.5 months, #7: 8.5 months, #8: 16 months, #9: 12 months, #10: 17.8 months.
Description: All AEs were collected and classified per CTCAE version 5.0. However, only those AEs and SAEs that were attributed by the investigators to be possibly, probably, or definitely related to FLASH radiotherapy were used for the assessment of toxicity of the FLASH treatment. There were no SAEs attributed to FLASH treatment, and the 7 AEs attributed to FLASH treatment were listed in the table as "Treatment Related". The remaining AEs in the table were unrelated to FLASH.
Arm/Group | FLASH Radiotherapy for Painful Bone Metastasis(-es)
All-Cause Mortality (participants affected / at risk) | 6/10
Serious Adverse Events (participants affected / at risk) | 7/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FLASH Radiotherapy for Painful Bone Metastasis(-es) (N=10)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1
Confusion (Psychiatric disorders) | 1
Disease Progression (General disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Fever (General disorders) | 1
Hepatic Failure (Hepatobiliary disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Lung Infection (Infections and infestations) | 3
Nausea (Gastrointestinal disorders) | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Disease (Cardiac disorders) | 1
Skin Infection (Skin and subcutaneous tissue disorders) | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FLASH Radiotherapy for Painful Bone Metastasis(-es) (N=10)
Treatment Related Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 4
Treatment Related Pruritis (Skin and subcutaneous tissue disorders) | 2
Treatment Related Edema limb (General disorders) | 1
Treatment Related Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Treatment Related Skin discoloration (Skin and subcutaneous tissue disorders) | 1
Treatment Related Fatigue (General disorders) | 1
Treatment Related Erythema (Skin and subcutaneous tissue disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Activated Partial Thromboplastin Time Prolonged (Investigations) | 3
Agitation (Psychiatric disorders) | 1
Akathisia (Nervous system disorders) | 1
Alanine aminotransferase increased (Investigations) | 4
Alkaline Phosphatase Increased (Investigations) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 3
Ankle fracture (Injury, poisoning and procedural complications) | 1
ANC Decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 4
Anxiety (Psychiatric disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Ascites (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 6
Blood Bicarbonate Decreased (Investigations) | 1
Blood bicarbonate Increased (Investigations) | 1
Blood Bilirubin Increased (Investigations) | 3
Blood Lactate Dehydrogenase Increased (Investigations) | 2
Blurred Vision (Eye disorders) | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 3
Cardiac Troponin Increased (Investigations) | 3
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 2
Chills (General disorders) | 2
Chronic Kidney Disease (Renal and urinary disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Concentration Impairment (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 4
Constipation (Gastrointestinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine Increased (Investigations) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Dental Caries (Gastrointestinal disorders) | 1
Depression (Psychiatric disorders) | 2
Diarrhea (Gastrointestinal disorders) | 4
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1
Dizziness (Nervous system disorders) | 2
Dry Mouth (Gastrointestinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Dysuria (Renal and urinary disorders) | 3
Ear Pain (Ear and labyrinth disorders) | 1
Edema Face (General disorders) | 2
Edema Limb (General disorders) | 3
Ejection Fraction Decreased (Investigations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Epstein-Barr Virus Infection (Infections and infestations) | 1
Eye Pain (Eye disorders) | 1
Facial Asymmetry (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Fatigue (General disorders) | 6
Fecal Incontinence (Gastrointestinal disorders) | 2
Fever (General disorders) | 2
Fibrinogen (Investigations) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Flu-like Symptoms (General disorders) | 2
Flushing (Vascular disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Gait Disturbance (General disorders) | 1
Gastroesophageal Reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders, other - mouth sores (Gastrointestinal disorders) | 2
General Disorders & Administration Site Conditions, other- Chest tightness (General disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 3
Hematoma (Perinephric) (Vascular disorders) | 1
Hematuria (Renal and urinary disorders) | 5
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 9
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hypotension (Vascular disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Ileus (Gastrointestinal disorders) | 1
Infections and infestations - Other, COVID-19 (Infections and infestations) | 2
Infections and infestations - Other, Strep throat (Infections and infestations) | 1
Injury, poisoning and procedural complications, other- Pain/injury to side (Injury, poisoning and procedural complications) | 1
INR Increased (Investigations) | 3
Insomnia (Psychiatric disorders) | 3
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1
Localized Edema (General disorders) | 2
Lung Infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 6
Malaise (General disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Morbilliform rash (Skin and subcutaneous tissue disorders) | 1
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness Upper Limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, clavical pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorders, other- Back weakness (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Neoplasms benign, malignant and unspecified - Other, Baker's Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neutrophil count decreased (Investigations) | 2
Nipple Deformity (Reproductive system and breast disorders) | 1
Non-cardiac Chest Pain (General disorders) | 1
Other - Erythema (left tibia) (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Other - Low Iron (Metabolism and nutrition disorders) | 1
Other - Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1
Other - unspecified rash (Skin and subcutaneous tissue disorders) | 2
other- Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Other - hip pain (Injury, poisoning and procedural complications) | 1
Other - Pulmonary embolism (Vascular disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2
Paresthesia (Nervous system disorders) | 1
Periorbital Edema (Eye disorders) | 2
Platelet count decreased (Investigations) | 6
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Presyncope (Nervous system disorders) | 1
Proteinuria (Renal and urinary disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Rectal Hemorrhage (Gastrointestinal disorders) | 1
Renal and urinary disorders, other- Azotemia (Renal and urinary disorders) | 1
Renal Calculi (Renal and urinary disorders) | 2
Renal Colic (Renal and urinary disorders) | 1
Reproductive System and Breast Disorders, other- Primary ovarian insufficiency (Reproductive system and breast disorders) | 1
Retinal Detachment (Eye disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 2
Skin and subcutaneous tissue disorders, other- Grey hair (Skin and subcutaneous tissue disorders) | 1
Skin infection (Skin and subcutaneous tissue disorders) | 1
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid Stimulating Hormone Increased (Investigations) | 1
Tremor (Nervous system disorders) | 1
Upper Respiratory Infection (Infections and infestations) | 1
Urinary Frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Urinary Urgency (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Watering Eyes (Eye disorders) | 1
Weight Gain (Investigations) | 3
Weight Loss (Investigations) | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
White Blood Cell Decreased (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT04592887/Prot_SAP_000.pdf